CLINICAL TRIAL: NCT06334328
Title: Feasibility and Acceptability of Virtual Reality-based Mindful Movement Therapy for Older Adults
Brief Title: Virtual Reality-based Mindful Movement Therapy for Seniors
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Drexel University (Other)
Responsible Party: Principal Investigator, Minjung Shim, PhD, Assistant Professor, Drexel University
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Other
Other Study IDs: 2205009237
Record Dates: First submitted 2022-07-29; First posted 2024-03-28 (Actual); Last update posted 2024-03-28 (Actual); Status verified 2024-03

CONDITIONS: Cognitive Decline; Physical Activity; Psychological Wellbeing
MeSH Terms: conditions — Cognitive Dysfunction; Motor Activity

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (1):
- Virtual reality based mindful movement therapy (Experimental): Participants will be asked to complete 12 VR-MMT sessions over a 6-week period, with two 30-minute sessions per week.
  Each session will be comprised of a guided warm-up (5 min, pre-recorded video played on the computer monitor) followed by a VR module with a head-mounted display (HMD) on (20 min). The VR module includes both structured and freestyle dance/movement guided by the therapist's prompts that are pre-recorded. Sessions will end with a closing routine (5 min, including guided breathing, stretching, and meditation) in order to assist participants to transition back to the real environment.
  Interventions: Behavioral: Virtual reality based mindful movement therapy

INTERVENTIONS:
Behavioral: Virtual reality based mindful movement therapy — VR-MMT combines VR games, multisensory and cognitive stimulation, hand-eye and full body coordination, creative processes, expressive movement, mindfulness practice, and social connectedness.

SUMMARY:
The current proposal aims to 1) develop a technical platform and implementation plan for the delivery of a virtual reality-based mindful movement therapy (VR-MMT) protocol for older adults; and 2) conduct a clinical trial to examine the feasibility and preliminary efficacy of an 8-week, 16-session module VR-MMT intervention for this population. The findings of this study will help us to identify engagement barriers and refine the intervention contents as well as the study protocol necessary for the preparation of grant applications to conduct a controlled clinical trial. This study is innovative and high impact as this is the first study to examine the feasibility and preliminary efficacy of a VR-MMT intervention that could potentially ameliorate cognitive and mobility decline and promote psychological wellbeing in older adults by combining a widely accessible technology and creative embodiment-based approach.

DETAILED DESCRIPTION:
Age-related cognitive decline is a significant public health issue. Despite the benefit of regular physical activity in preserving cognitive function and overall health and wellbeing, approximately 30% of older adults are physically inactive due to a lack of motivation and other engagement barriers. Further, social isolation and loneliness are common in older adults which are associated with an increased risk of developing Alzheimer's disease (AD) and dementia. A combination of physical and cognitive training appears to be effective to improve cognitive function in older adults experiencing cognitive deterioration. Growing evidence suggests virtual reality(VR) is a promising tool to improve cognitive functioning in older adults. We have developed a novel virtual reality-based mindful movement therapy (VR-MMT) program for older adults that combines VR games, multisensory and cognitive stimulation, hand-eye and full body coordination, creative processes, expressive movement, mindfulness practice, and social connectedness. The current proposal aims to 1) develop a technical platform and implementation plan for the delivery of a VR-MMT protocol for older adults; and 2) conduct a clinical trial to examine the feasibility and preliminary efficacy of an 8-week, 16-session module VR-MMT intervention for this population. The findings of this study will help us to identify engagement barriers and refine the intervention contents as well as the study protocol necessary for the preparation of grant applications to conduct a controlled clinical trial. As this is the first study to examine the feasibility and preliminary efficacy of a VR-MMT intervention that could potentially ameliorate cognitive and mobility decline and promote psychological wellbeing in older adults by combining a widely accessible technology and creative embodiment-based approach, it meets the definition of "innovative, high impact" research. Our specific aims include:

Aim 1: To develop (a) a technical platform and (b) an implementation plan for the delivery of a VR-MMT intervention for older adults. Technical development and implementation planning will be guided by the expert project team with key input from community stakeholders.

Aim 2: To conduct a clinical feasibility trial to examine the safety, feasibility, and preliminary efficacy (primary outcomes: cognitive function, psychological wellbeing, physical activity participation, secondary outcomes: mobility performance, loneliness, self-efficacy) of an 8-week VR-MMT intervention for older adults.

ELIGIBILITY:
Inclusion Criteria:

* Subjects must be age 65 or older at the time of informed consent.
* Able to move and stand without assistance
* Subjects must be proficient in spoken and written English for consenting as well as for study participation
* Subjects with medical conditions must be stable for these conditions. Stable control on medication is acceptable.
* Subject must have normal visual acuity (or corrected to normal) and normal color vision as indicated by self-report.
* Subject must have adequate hearing acuity as indicated by self-report.

Exclusion Criteria:

* Existing diagnosis of a neurodegenerative disorder (e.g., Alzheimer's Disease, Lewy Body Dementia, Frontal-Temporal Dementia).
* Prior diagnosis that might impact cognition and movement abilities including: cardiovascular or respiratory illness or injury, substance abuse, schizophrenia, bipolar disorder, or other neurological diseases (e.g., epilepsy, Parkinson's disease, seizure disorder).
* Affirmative answer to any Physical Activity Readiness Questionnaire for 70+ year-old adults (PAR-Q-70+) questionnaire.

Min Age: 65 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Older Adult
Enrollment: 12 (Actual)
Dates: Start 2022-08-15 (Actual); Primary Completion 2023-09-30 (Actual); Study Completion 2024-01-31 (Actual)

PRIMARY OUTCOMES:
Treatment adherence | Throughout the intervention (week 1-week 6)
  We will log participants' session attendance to track treatment adherence
Treatment acceptability | Post intervention (Week 6)
  Treatment Evaluation Inventory Short Form (post-intervention only) is a 9-item measure of the perceived acceptability of behavioral treatments. Items are rated on a 5-point scale with the anchor points 1 (strongly disagree) and 5 (strongly agree). Higher score meaning greater levels of treatment acceptability.
Treatment satisfaction | Post intervention (Week 6)
  Usefulness, Satisfaction, and Ease of Use Questionnaire (post-intervention only) is a 30-item instrument that examines four dimensions of usability: usefulness, ease of use, ease of learning, and satisfaction. Each question is rated on a seven-point scale with the anchor points 1 (strongly disagree) and 7 (strongly agree). There are also two open-ended response questions asking the user to list the most negative aspects and the most positive aspects. All items are summed to give a total score, with higher scores indicating greater usability.
Qualitative feedback | Post intervention (within 1-2 weeks after the conclusion of the 6-week intervention)
  A semi-guided individual interview (30 min) will be conducted upon the completion of the intervention to learn about participants' experience of participating in the study, perceived benefits, perceived barriers, and suggestions for improvement.
Safety | Throughout the intervention (week 1-week 6)
  We will log adverse event to assess safety of the intervention

SECONDARY OUTCOMES:
Montreal Cognitive Assessment (MoCA) | Pre and post intervention (Week 0 and Week 6)
  MoCA assesses different cognitive domains: attention and concentration, executive functions, memory, language, conceptual thinking, calculations, and orientation.
Trail making test | Pre and post intervention(Week 0 and Week 6)
  Trail-Making Test is a measure of attention, speed, and mental flexibility. It also tests spatial organization, visual pursuits, recall, and recognition.
The Warwick-Edinburgh Mental Well-being Scale (WEMWBS) | Pre and post intervention(Week 0 and Week 6)
  WEMWBS is a 14-item scale of mental well-being covering subjective well-being and psychological functioning, in which all items are worded positively and address aspects of positive mental health.
Physical Activity Scale for the Elderly (PASE) | Pre and post intervention(Week 0 and Week 6)
  PASE is a 10-item scale that uses frequency, duration, and intensity level of activity over the previous week to assign a score, ranging from 0 - 793, with higher scores indicating greater physical activity.
Physical Performance Battery (SPPB) | Pre and post intervention(Week 0 and Week 6)
  SPPB will be administered to assess mobility performance. SPPB is a group of measures that combines the results of gait speed, chair stand, and balance tests developed using data from a large population-based epidemiologic study of older persons. It consists of repeated chair stands, balance testing, and walking.
General Self-Efficacy Scale | Pre and post intervention(Week 0 and Week 6)
  General Self-Efficacy Scale is a 10-item scale measuring self-efficacy, which has been correlated with positive emotion, optimism, and work satisfaction.
Positive Affect and Negative Affect Scale (PANAS) | Pre and post intervention(Week 0 and Week 6)
  PANAS is a 20-item self-report measure of affect. The total score is calculated by finding the sum of the 10 positive items and the 10 negative items.

CONTACTS AND LOCATIONS:
Locations (1):
- Drexel Universitsy, Philadelphia, Pennsylvania, United States

IPD SHARING:
Plan to Share IPD: No